CLINICAL TRIAL: NCT03280524
Title: Reflexology and Quality of Life in Diabetic Patients
Brief Title: Reflexology and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, Beatriz Bertolaccini Martínez, Professor, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CAAE: 30795814.8.0000.5102
Record Dates: First submitted 2017-09-07; First posted 2017-09-12 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2017-09

CONDITIONS: Diabetic Foot
Keywords: Reflexology,diabetes, quality of life
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus | interventions — Musculoskeletal Manipulations; Massage; Educational Status

STUDY DESIGN:
Intervention Model Description: The patients will be taken to a room reserved for the procedure. First, the patients answer the research instruments and then they will be asked to lie supine on a stretcher. The feet of the patients will be cleaned with water (37ºC) and mild soap and then will be dry with paper towels. The next phase consists in the application of foot massage, that will follow the Lourenço's Protocol (2012), which consists of 14 steps of relaxation massage. Each step will have duration of 1 minute, 3 procedures by week, by 4 consecutive weeks. The research instruments, SF-36 and Stanford Health Assessment Questionnarie will be applied before the first and after the last procedure.
Who Masked: Participant, Investigator
Masking Description: To ensure the blinding, the study included an interventionist enabled for application of foot reflexology.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Control Group will receive self-care guidelines with feet
  Interventions: Other: self-care guidelines with feet
- Treatment Group (Experimental): Treatment will receive self-care guidelines with feet and 12 sessions of foot reflexology
  Interventions: Other: reflexology; Other: self-care guidelines with feet

INTERVENTIONS:
Other: reflexology
  Other Names: massage
  Arms: Treatment Group
Other: self-care guidelines with feet
  Other Names: education

SUMMARY:
This is a randomized, controlled and blind clinical trial with 60 type 2 diabetes patients divided into 2 groups of 30 patients each, Control Group (CG) and Treatment Group (TG). The TG will receive self-care guidelines with feet and 12 sessions of foot reflexology, while the CG will only receive the guideline.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effects of reflexology on the quality of life and functional capacity of patients at risk for diabetic neuropathy. This is a randomized, controlled and blind clinical trial with type 2 diabetes patients. The eligibility criteria are 10 years or more of diagnosis of diabetes mellitus, between the ages of 50 to 75 years, both sexes, and registered in the Primary Health Care Unit of São João or in the Diabetes Education Center in Minas Gerais state, Brazil. As exclusion criteria, it will be considered the presence of ulcers in the feet, amputations of the lower limbs, deficits in cognitive abilities, and previous treatment using reflexology. For the calculation of the sample size, a pilot test will be conducted with 8 diabetic patients. It will be used the statistical software Biostat® 5.3. The sample found was of 60 patients who were divided into 2 groups of 30 patients each, Control Group (CG) and Treatment Group (TG). The TG will receive self-care guidelines with feet and 12 sessions of foot reflexology, while the CG will only receive the guideline. For the evaluations, it will be applied the instrument for quality of life (SF-36) and for functional capacity, the Stanford Health Assessment Questionnaire. This research will follow the standards set by resolution 466/12 of the National Health Council, for research with human beings and will be conducted in accordance with the ethical recommendations of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* 10 years or more of diagnosis of diabetes mellitus, between the ages of 50 to 75 years, both sexes, and registered in the Primary Health Care Unit of São João or in the Diabetes Education Center in Minas Gerais state, Brazil.

Exclusion Criteria:

* presence of ulcers in the feet, amputations of the lower limbs, deficits in cognitive abilities, and previous treatment using reflexology

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Quality of Life Questionnaire SF-36 | An average of 1 year
  measure of quality of life

OTHER OUTCOMES:
Stanford Health Assessment Questionnaire | An average of 1 year
  measure of functional capacity

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Ms Martínez, doctor, Principal Investigator — Universidade do Vale do Sapucai
Locations (1):
- Diabetes Education Center, Pouso Alegre, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aguiar CC, Vieira AP, Carvalho AF, Montenegro-Junior RM. [Assessment instruments for a Health-Related Quality of Life in diabetes mellitus]. Arq Bras Endocrinol Metabol. 2008 Aug;52(6):931-9. doi: 10.1590/s0004-27302008000600004. Portuguese. PMID 18820804
- [Background] Kaul K, Tarr JM, Ahmad SI, Kohner EM, Chibber R. Introduction to diabetes mellitus. Adv Exp Med Biol. 2012;771:1-11. doi: 10.1007/978-1-4614-5441-0_1. PMID 23393665
- [Background] Tiran D, Chummun H. The physiological basis of reflexology and its use as a potential diagnostic tool. Complement Ther Clin Pract. 2005 Feb;11(1):58-64. doi: 10.1016/j.ctnm.2004.07.007. PMID 15984227
- [Background] Armstrong AR, Thiebaut SP, Brown LJ, Nepal B. Australian adults use complementary and alternative medicine in the treatment of chronic illness: a national study. Aust N Z J Public Health. 2011 Aug;35(4):384-90. doi: 10.1111/j.1753-6405.2011.00745.x. PMID 21806735
- [Background] Wang MY, Tsai PS, Lee PH, Chang WY, Yang CM. The efficacy of reflexology: systematic review. J Adv Nurs. 2008 Jun;62(5):512-20. doi: 10.1111/j.1365-2648.2008.04606.x. PMID 18489444
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366